CLINICAL TRIAL: NCT03473067
Title: Community Level Primary Prevention of Dating and Sexual Violence in Middle Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lifespan (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Lindsay Orchowski Ph.D., Staff Psychologist, Lifespan
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1U01CE002651 (NIH)
Record Dates: First submitted 2017-08-28; First posted 2018-03-22 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Violence
MeSH Terms: interventions — Capacity Building

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Norms Marketing (Experimental): This arm includes a social norms marketing campaign tailored to the school.
  Interventions: Behavioral: Social Norms Marketing Campaign
- Capacity Building (Active Comparator): This arm includes a series of teacher training, and parent engagement meetings, with the goal of building capacity to address violence in the school.
  Interventions: Other: Capacity Building

INTERVENTIONS:
Behavioral: Social Norms Marketing Campaign — This poster based marketing campaign is designed to correct inaccurate perceptions of norms regarding violence.
  Other Names: Your Voice Your Data
  Arms: Social Norms Marketing
Other: Capacity Building — Schools will participate in teacher training and parent training.
  Arms: Capacity Building

SUMMARY:
Dating and sexual violence are significant public health concerns occurring on a continuum of severity across the lifespan, with serious consequences to victims and society. The present research advances the science of prevention by rigorously evaluating a comprehensive social norms marketing campaign to promote community-level change in dating and sexual violence in middle schools. Partnership between researchers and a CDC Rape Prevention and Education Program (RPE) funded agency is a core feature of this work, and aims to build community capacity to implement and evaluate violence prevention efforts, and promote the subsequent uptake of social norms marketing campaigns as a strategy for reducing dating and sexual violence among youth.

DETAILED DESCRIPTION:
In a group cluster trial, a comprehensive, tailored, data-based social norms marketing campaign that addresses misperceptions of: 1) the acceptability of dating and sexual violence; 2) gender roles; 3) sexual activity; 4) sexual communication/consent; 5) support for victims; and 6) bystander intervention will be evaluated among middle schools. Poster messaging will be paired with several systematic efforts to diffuse program content through the community, including a Lunch and Learn Teacher Training, Social Norms Video, Teacher Workbook, Parent Mailing, and Parent Information Session. A member of the researcher-practitioner team, designated as a School Resource Provider, will oversee campaign implementation in partnership with a teacher champion. The Resource Provider will also track campaign intensity, assess campaign credibility through intercept interviews with teachers and students, work with teachers to infuse messaging into classroom activities, and assist the teacher champion with addressing "kick-back" to the campaign. Outcome assessments will be completed by teachers, administrators and students. Towards the goal of exploring the role of other environmental factors as moderators of program effects, school administrators will assess their community readiness to develop and implement school dating and sexual violence prevention policy, in general, and social norms marketing, in particular. A neighborhood scan will also be conducted to estimate the density of nearby outlets associated with gender-based personal violence.

ELIGIBILITY:
Inclusion Criteria:

* Student at a middle school or teacher/administrator at a middle school
* Provide student assent and parental consent as specified in protocol or provide adult consent for study participation

Exclusion Criteria:

• None

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4344 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Sexual Violence Victimization | Over 6 months
  Rates of sexual violence victimization
Dating Violence Victimization | Over 6 months
  Rates of dating violence victimization
Sexual Violence Perpetration | Over 6 months
  Rates of sexual violence perpetration
Dating Violence Perpetration | Over 6 months
  Rates of dating violence perpeptration

SECONDARY OUTCOMES:
Bystander Intervention | Over 6 months
  Rates of bystander intervention
Attitudes Towards Violence | Change from baseline to 6 months
  Attitudes towards violence scale

OTHER OUTCOMES:
Teacher Engagement in Bystander Intervention | Over 6 months
  Rates of bystander intervention behavior among teachers
Perceptions of Social Norms | Change from baseline to 6 months
  A series of items were developed for the purpose of the present study to assess student perceptions of peer norms regarding dating and sexual violence. Items are scored on a range of 0% - 100% to indicate the percent of peers within the school that would endorse each item. Scores for each item will be examined individually. Positive scores on this measure are indicated when respondents perceive a greater number of their peers would endorse healthy behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay M. Orchowski, Ph.D., Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No